CLINICAL TRIAL: NCT05652803
Title: Bibliotherapy-based Psychoeducation Program the Effect of Elderly Individuals on Depression and Hopelessness Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Esra Bekircan, PhD student, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: bibliotherapy
Record Dates: First submitted 2022-12-02; First posted 2022-12-15 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Elderly People; Depressive Symptoms; Despondency
Keywords: Bibliotherapy; elderly individuals; depression; despair; psychoeducation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: This research is a randomized controlled experimental study to compare the effects of two psychoeducational programs prepared in accordance with the principles of psychoeducation and bibliotherapy on the depression and hopelessness levels of elderly individuals. In this study, there are pre-test, post-test, follow-up test and comparative experimental group. In this model, there are 2 different experimental groups and 1 control group created by randomization. No intervention will be made in the control group. There will be 13 people in each group.
Who Masked: Investigator
Masking Description: In this study, simple random sampling method was used, in which individuals were selected as samples using probability rules. When using the simple random sampling method, the units in the universe are listed and numbered first. Then, the elements to be included in the sample are determined by using the "Draw Method" or "Random Numbers Table". 39 people who accepted to participate in this study and met the inclusion criteria were assigned to the experimental and control groups by simple randomization method. In order to reduce the selection bias, while determining the experimental and control groups, the assignment of the experimental and control groups by the randomization method from the random numbers table by a statistician who did not have a direct role in the research (https://www.random.org/integers/ random numbers table). group: 13, 2nd experimental group: 13, control group: 13).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bibliotherapy-based psychoeducation program (Experimental): In the bibliotherapy-based psychoeducation program sessions, techniques such as information and discussion based on the bibliotherapy method were included. Brief information will be given for 5-10 minutes in each session. At the end of the sessions, exercises will be given to reinforce the knowledge and skills acquired by the group members in the sessions and to transfer them to daily life, and the sessions will be concluded.
  Interventions: Behavioral: bibliotherapy-based psychoeducation program
- Psychoeducation Program (Experimental): The General Purpose of the Psychoeducation Program for Reducing Depression and Hopelessness: To help the participants gain awareness, skills and attitudes in order to help them reduce their depression and hopelessness levels.
  Interventions: Behavioral: psychoeducation program

INTERVENTIONS:
Behavioral: bibliotherapy-based psychoeducation program — In this study, the researcher aimed to gain awareness, skills and attitudes in order to help the participants reduce the negative consequences of depression and hopelessness. Based on the general purpose, a separate target has been established for each session of both intervention types. For bibliotherapy-based psychoeducation, story texts compatible with the goals were added to each session, and the psychoeducation part was supported by bibliotherapy. Considering the ability of the elderly to attend the training regularly, their attention and coordination, it was decided that the study would consist of 6 sessions and each session would be 60 minutes on average.
  Arms: bibliotherapy-based psychoeducation program
Behavioral: psychoeducation program — The General Purpose of the Psychoeducation Program for Reducing Depression and Hopelessness: To help the participants gain awareness, skills and attitudes in order to help them reduce their depression and hopelessness levels.
  Arms: Psychoeducation Program

SUMMARY:
Bibliotherapy has been mainly focused on the social and emotional problems of children and young people, and studies with the elderly are very few. Based on the suggestion of meeting the right book with the right individual, which is the basis of bibliotherapy, it is predicted that the bibliotherapy method can be useful in reducing depression and increasing hope in the elderly, with the selection of books that are suitable for the cognitive levels of the elderly.

DETAILED DESCRIPTION:
Today, one of the most important social changes is the aging of the world population. The number and rate of elderly individuals is increasing in the populations of almost all countries in the world. During the aging process, increasing number and severity of health problems, decreasing functional abilities, loss of spouse and friends, financial constraints, retirement, loss of social status are the problems that elderly individuals can potentially encounter in life change. In the face of these problems, the elderly may feel worthless and experience negative feelings such as depression and hopelessness.

Nurses have important responsibilities in the health services provided to elderly individuals in the old age, when hopelessness and depression can be experienced intensely. Cognitive and mental status are considered in the evaluation of the elderly individual. In this sense, in the approach to the elderly person with depression, the nurse should make a comprehensive assessment of the signs and symptoms of depression that may be seen in the individual. The aim of nursing care includes taking a role in the prevention, recognition, treatment and care of depression. The more effective use of the independent roles of the nurse in nursing care increases the quality of the care provided. One of the methods to be applied in this sense is art therapy.

Art therapy is a supportive treatment method that enables individuals to express themselves, gain coping skills and increase their resilience by using art as a tool in the Nursing Intervention Classification. It helps them to develop their interpersonal skills, reduce stress, manage their behavior, increase their self-esteem, self-confidence and gain insight.Creating art and reflecting it on art products can increase individuals' self-confidence, enable them to cope with stress and other traumatic experiences, improve their cognitive skills and enjoy life.

Bibliotherapy, which can be expressed as a method of improving mental health through reading, includes the use of non-fiction self-help books, as well as the treatment of emotional and behavioral disorders through a literary work, poem or film. As a matter of fact, studies have shown that tales, stories and myths are effective tools in counseling and contribute to the healing of clients. This technique has been used successfully in the treatment of many problems in children, adolescents, adults and the elderly and its effectiveness has been proven. Bibliotherapy has been mainly focused on the social and emotional problems of children and young people, and studies with the elderly are very few. Based on the suggestion of meeting the right book with the right individual, which is the basis of bibliotherapy, it is predicted that the bibliotherapy method can be useful in reducing depression and increasing hope in the elderly, with the selection of books that are suitable for the cognitive levels of the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years or older
* A score between 5 and 11 on the Geriatric Depression scale (mild to moderate)
* Not having a perception disorder that will prevent communication
* Volunteering to participate in the research

Exclusion Criteria:

* • Having a communication barrier,

  * Having been diagnosed with dementia,
  * Being diagnosed with a severe psychiatric illness
  * Having a terminal illness

Exclusion Criteria:

* Not attending any session of the six-session training program and not attending the make-up session,
* Not participating in any of the Pretest, Posttest- and Follow-up tests.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
geriatric depression | 6 weeks
  In line with the training given, it is aimed to decrease the level of geriatric depression.

SECONDARY OUTCOMES:
despair | 6 weeks
  In line with the education given, it is aimed to decrease the hopelessness level of the elderly individuals.

CONTACTS AND LOCATIONS:
Overall Officials: ayşe okanlı, Study Director — a.okanliægmail.com
Locations (1):
- Trabzon Retirement Association, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
1. Experimental Group--Bibliotherapy-based psychoeducation program (6 sessions)
  2. Experimental Group-- psychoeducation program (6 sessions) control group--no intervention
Time Frame: After the pretest applied by the researcher to the 1st experimental group, 2nd experimental group and control group, psychoeducational programs, which are the independent variables in this research, will be applied to the 1st and 2nd experimental groups. After this application, post-test and follow-up tests will be given to all three groups and the effectiveness of psychoeducation programs will be compared.

REFERENCES:
- See also: Effects of Developmental Bibliotherapy on Subjective Well-Being of Older Adults Living in Nursing Homes: A Quasi-Experimental Study — https://pubmed.ncbi.nlm.nih.gov/35191766/
- See also: Culture Change in Nursing Homes: What Is the Role of Nursing Home Resources? — https://pubmed.ncbi.nlm.nih.gov/30015532/
- See also: How effective is bibliotherapy for very old adults with subthreshold depression? A randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/20808151/
- See also: The effectiveness of a bibliotherapy in increasing the self-management ability of slightly to moderately frail older people. — https://pubmed.ncbi.nlm.nih.gov/15939567/